CLINICAL TRIAL: NCT00815841
Title: Methylphenidate in Healthy Young Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: VARDA GROSS-TSUR MD, SHAARE ZEDEK MEDICAL CENTER
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ShaareZMC.ctil
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Healthy
Keywords: Determine the effect of MPH on a diagnostic continuous performance task that assesses attention and on a decision making test in young healthy adults
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: METHYLPHENIDATE — 15-20mg during one of the two sessions

SUMMARY:
Background: There is a paucity of data as to the effect of methylphenidate (MPH) on young adults who do not have attention deficit hyperactivity disorder (ADHD). The existing data is equivocal and focuses on neuropsychological functions that are not always relevant to the clinical aspects of attention. Objective: To determine the effect of MPH on a diagnostic continuous performance task that assesses attention per se (TOVA) and on a decision making test (Modified Gamble Decision Test) in young, healthy adults. Methods: Fifty young adults, men and women ages 20-30, without ADHD, learning disabilities, history of past or present use of MPH or other psychotropic drugs, will be eligible to participate. Design: The experiment will be conducted in 2 sessions, the first lasting 3.5 hours and the second 2.5 hours in a randomized, double-blind prospective design. In the first session, the subjects will be screened for ADHD past and present, major psychiatric diagnosis (depression, anxiety, etc), use of MPH in the past, psychotropic medications or recreational drugs and any other chronic illness; urine will be tested for beta-hCG to rule out pregnancy. Blood pressure and heart rate will be measured. The participants will then be given either placebo or MPH (15-20 mg) and after 90 minutes will proceed to complete the TOVA (that lasts 22 minutes) and Modified Gamble-Decision Test (15 minutes). Before taking the pill and prior to the testing, the subjects will complete the Visual Analogue Scale (VAS) which quantifies their subjective feelings regarding present mental and emotional state. In the second session, 2 weeks later, blood pressure and heart will be measured and the VAS completed prior to and 90 minutes after taking the tablet. The subjects then undergo the TOVA and Modified Gamble-Decision Test. Data Analysis: will be performed using the paired t-tests for parametric variables and one way ANOVA with repeated measurements. Significance: Results of this study are important since MPH is used and abused by healthy students as a "study aid" although its objective effects in normal young adults are not well delineated

ELIGIBILITY:
Inclusion Criteria:

* ages 20-30

Exclusion Criteria:

* ADHD
* learning disabilities
* history of past or present use of MPH or other psychotropic drugs
* pregnancy
* chronic illness

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The TOVA score | January - December 2009